CLINICAL TRIAL: NCT05148169
Title: A Pilot Study on Effect of add-on Sulforaphane to SSRIs and Application of Niacin Skin Flush Response Test in Major Depressive Disorder
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201940109
Record Dates: First submitted 2021-12-02; First posted 2021-12-08 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-11

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; Sulforaphane; Niacin skin flush response; Marker; Add-on
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Selective Serotonin Reuptake Inhibitors; sulforaphane

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SSRI group (Active Comparator): One SSRI is prescribed based on treatment guidelines for major depressive disorder and drug prescription manual. The dose is 20-60mg/day for fluoxetine, 20-40mg/day for paroxetine, 100-300mg/day for fluvoxamine, 50-200mg/day for sertraline, 20-40mg/day for citalopram, 10-20mg/day for escitalopram, respectively.
  Interventions: Drug: SSRIs
- SSRI plus Sulforaphane group (Experimental): One SSRI is prescribed based on treatment guidelines for major depressive disorder and drug prescription manual. The dose is 20-60mg/day for fluoxetine, 20-40mg/day for paroxetine, 100-300mg/day for fluvoxamine, 50-200mg/day for sertraline, 20-40mg/day for citalopram, 10-20mg/day for escitalopram, respectively.
  The oral dose of SFN is based on weight. The usage and dosage are as follows: 40-70kg, 4 tablets/day (containing 274μmol of glucosinolates); 70-90kg, 6 tablets/day (containing 411μmol of glucosinolates). Take it once in the morning and evening.
  Interventions: Drug: SSRIs; Dietary Supplement: SSRI plus Sulforaphane
- Healthy control group (No Intervention): No intervention is given.

INTERVENTIONS:
Drug: SSRIs — One SSRI(No-specified) is prescribed based on treatment guidelines for major depressive disorder and drug prescription manual. The dose is 20-60mg/day for fluoxetine, 20-40mg/day for paroxetine, 100-300mg/day for fluvoxamine, 50-200mg/day for sertraline, 20-40mg/day for citalopram, 10-20mg/day for escitalopram, respectively.
  Arms: SSRI group; SSRI plus Sulforaphane group
Dietary Supplement: SSRI plus Sulforaphane — One SSRI(No-specified) is prescribed based on treatment guidelines for major depressive disorder and drug prescription manual. The dose is 20-60mg/day for fluoxetine, 20-40mg/day for paroxetine, 100-300mg/day for fluvoxamine, 50-200mg/day for sertraline, 20-40mg/day for citalopram, 10-20mg/day for escitalopram, respectively.
  The oral dose of SFN (ZHIYINGUOSU, Shenzhen Fushan Biotech Co. Ltd.) is based on weight. The usage and dosage are as follows: 40-70kg, 4 tablets/day (containing 274μmol of glucosinolates); 70-90kg, 6 tablets/day (containing 411μmol of glucosinolates). Take it once in the morning and evening.
  Arms: SSRI plus Sulforaphane group

SUMMARY:
A 12-week, randomized controlled trial (RCT) will be conducted to explore the effect of add-on sulforaphane (SFN) to selective serotonin reuptake inhibitors (SSRIs) for major depressive disorder (MDD). This study also aims to explore the value of niacin skin flush response test in MDD. One hundred adults diagnosed with MDD will be recruited. Then all the patients will be randomly assigned to SSRI only group and SSRI plus SFN group. Clinical symptoms and side-effects will be evaluated using the 17-Hamilton Depression Rating Scale (17-HDRS), the Hamilton Anxiety Scale (HAMA), Treatment Emergent Symptom Scale (TESS), and Asberg's Rating Scale for Side Effects (SERS) at baseline and weeks 2, 4, 8 and 12 after treatment. Fifty healthy subjects will be recruited as control group. For all subjects, testing of niacin skin flush response and serum levels of nuclear factor erythroid-2-related factor 2(Nrf-2), p-Nrf2, Heme Oxygenase-1 (HO-1), malondialdehyde (MDA) and erythrocyte glutathion peroxidase (GPX) will be performed at baseline and endpoint. The primary outcome is the reduction rate in 17-HDRS total score from baseline to the end of the study. The secondary outcomes include changes in niacin skin flush response test and levels of serum markers. All the data will be analyzed by SPSS software.

ELIGIBILITY:
Inclusion Criteria:

1. aged 18-60 years;
2. diagnosed with moderate or severe depressive disorder according to the criteria of the DSM-5;
3. total score of 17-HDRS≥17;
4. never receiving electroconvulsive therapy (ECT)/modified ECT (MECT)/rTMS or other treatments in the past month;
5. having sufficient audio-visual ability and comprehension;
6. signed informed consent statements.

Exclusion Criteria:

1. serious or active somatic illness (abnormal index values were more than twice the limit of normal);
2. a history of mania/hypomania;
3. current high risk of suicide (score of item 3 of 17-HDRS ≥ 3);
4. pregnant or lactating women, or planning pregnant women;
5. taking immunosuppressants or vitamins recently.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
the reduction rate in 17-HDRS total score from baseline to the end of the study | at baseline, week 2/4/8/12 after treatment
  Remission is defined as 17-HDRS total score ≤7; Response is defined as ≥50% decrease from 17-HDRS total score at baseline and 17-HDRS total score>7; Nonresponse is defined as having a reduction of<50% on the total score of 17-HDRS comparing with baseline.
  at baseline, week 2/4/8/12 after treatment.

SECONDARY OUTCOMES:
changes in levels of serum markers from baseline to the end of the study | at baseline, week 8-12 after treatment
  changes in levels of serum markers including nuclear factor erythroid-2-related factor 2(Nrf-2), p-Nrf2, Heme Oxygenase-1 (HO-1), malondialdehyde (MDA) and erythrocyte glutathion peroxidase (GPX) from baseline to week 8-12 after treatment
changes in niacin skin flush response test from baseline to the end of the study | at baseline, week 8-12 after treatment
  changes in signals of blood flow (typified by maximum blood flow, MBF) detected by the Doppler Laser Flowmetry during the niacin skin flush response test from baseline to week 8-12 after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Mental Health Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided